CLINICAL TRIAL: NCT03520478
Title: A Phase III, Multicenter, Randomized, Open Study of SHR3680 Compared to Bicalutamide in the Treatment of Patients With Hormone Sensitive Prostate Cancer
Brief Title: A Study of SHR3680 in Treating Patients With Hormone Sensitive Prostate Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-3680-III-HSPC
Record Dates: First submitted 2018-04-27; First posted 2018-05-09 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer; Hormone-Dependent Prostate Cancer
Keywords: Hormone sensitive prostate cancer; SHR3680; Anti-androgen receptor
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SHR3680 (Experimental): Participants will receive SHR3680 orally
  Interventions: Drug: SHR3680
- bicalutamide (Active Comparator): Participants will receive bicalutamide orally
  Interventions: Drug: Bicalutamide

INTERVENTIONS:
Drug: SHR3680 — Tablet. Specifications of 80 mg; orally, once a day
  Arms: SHR3680
Drug: Bicalutamide — Tablet. Specifications of 50 mg; orally, once a day
  Arms: bicalutamide

SUMMARY:
The aim of this study is to compare the safety and efficacy of SHR3680 with bicalutamide in the treatment of patients with hormone sensitive prostate cancer.

DETAILED DESCRIPTION:
This is an open, multicenter, randomized phase III trial. This clinical study compares the efficacy and safety of SHR3680 with bicalutamide in the patients with hormone sensitive prostate cancer. Approximately 572 patients who meet the entry criteria will be randomly assigned in a 1:1 ratio to SHR3680 or bicalutamide treatment. Primary endpoints of the study are radiological progress-free survival (rPFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Age≧18 year, male;
* ECOG performance scale 0 to 1;
* Histologically or cytological confirmed prostate adenocarcinoma without neuroendocrine differentiation or small cell features ;
* Adequate hepatic, renal, heart, and hematological functions;
* Patients have given voluntary written informed consent before performance of any study-related procedure not part of normal medical care,with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Subject has received any prior radiation therapy or surgery for prostate cancer, except 1 course of palliative surgical therapy if it was used at least 4 weeks prior to day 1;
* Previous use or are using a second-generation androgen receptor antagonist (enzalutamide, ARN-509, ODM-201), abiraterone, ketoconazole for prostate cancer, or other agents that will inhibit the production of androgens;
* Have participated in an interventional clinical trial or been treated with the following drugs in the past 4 weeks prior to day 1: 5-alpha reductase inhibitors, estrogen, progestin, and herbal products known to decrease PSA levels ;
* Evidence of brain metastasis or primary tumors;
* Planned to initiate any other anti-tumor therapies during the study;
* Unable to swallow, chronic diarrhea and intestinal obstruction, or the presence of a variety of other factors that affect drug use and absorption; Clinically significant cardiovascular diseases;
* History of seizure or certain conditions that may predispose to seizure;
* Severe concurrent disease and infection that, in the judgment of the investigator, would make the patient inappropriate for enrollment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
rPFS | Approximately 70 months
  Time from randomisation to radiologically confirmed progressive disease or death due to any cause
OS | Approximately 70 months
  Time from randomisation to death due to any cause

SECONDARY OUTCOMES:
Time to prostate specific antigen (PSA) progression | Approximately 70 months
  Time from randomisation to the first time of PSA progression according to the criterion of PCGW3
Time to skeletal-related events | Approximately 70 months
  Time from randomisation to the first occurrence of a fracture or treatment for the fracture. The skeletal-related event is defined as the occurrence of either pathological or clinical fracture, spinal cord compression, bone-related radiotherapy or surgery
Objective response rate (ORR) | Approximately 70 months
  The percentage of subjects with measureable disease at baseline who achieved a complete or partial response in their soft tissue disease using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria
Time to initiation of a new antineoplastic therapy | Approximately 70 months
  Time from randomisation to the initiation of antineoplastic subsequent to the study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, M.D., Principal Investigator — Fudan University
Locations (67):
- Bulgaria (7):
  - Complex oncological center - Bourgas, Burgas
  - UMHAT 'Deva Maria'. EOOD, Burgas
  - MHAT - Dobrich. AD, Dobrich
  - MHAT 'Dr. Tota Venkova'. AD, Gabrovo
  - Complex Oncological Center - Plovdiv. EOOD, Plovdiv
  - MHAT 'Central Onco Hospital'. OOD, Plovdiv
  - Acibadem City Clinic Tokuda Hospital Ead, Sofia
- China (49):
  - Affiliated Hospital of Hebei University, Baoding
  - Beijing Cancer Hospital, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The third hospital of Peking University, Beijing
  - Tumor Hospital of the Chinese Academy of Medical Sciences, Beijing
  - China Japan Friendship Hospital of Jilin University, Changchun
  - The first hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Army characteristic medical center of the Chinese people's Liberation Army, Chongqing
  - Chongqing Cancer Hospital, Chongqing
  - The First Affiliated Hospital of Army Medical University, Chongqing
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Sun Yat-Sen hospital of Sun Yat-Sen University, Guangzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital of Zhejiang University Medicine college, Hangzhou
  - The Second affiliated hospital of zhejiang university medical college, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Zhejiang Province People's Hospital, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Qilu Hospital of Shandong University, Jinan
  - Yunnan Provincial Cancer Hospital, Kunming
  - The second hospital of Lanzhou University, Lanzhou
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Gulou Hospital Affiliated to Medical College of Nanjing University, Nanjing
  - Jiangsu Provincial Cancer Hospital, Nanjing
  - Jiangsu Provincial People's Hospital, Nanjing
  - Huadong Hospital of Fudan University, Shanghai
  - Ruijin Hospital, Shanghai
  - Shanghai General Hospital, Shanghai
  - The Cancer Hospital of Fudan University, Shanghai
  - Zhongshan Hospital of Fudan University, Shanghai
  - Liaoning Provincial Cancer Hospital, Shenyang
  - The fourth hospital of Hebei Medical University, Shijia Zhuang
  - The second hospital of Tianjin Medical University, Tianjing
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Hubei Provincial Cancer Hospital, Wuhan
  - Tongji Hospital, Tongji medical college of HUST, Wuhan
  - Union Hospital, Tongji Medical college of HUST, Wuhan
  - Wuxi People's Hospital, Wuxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Jiangsu Subei people's Hospital, Yangzhou
  - Henan people's Hospital, Zhengzhou
  - Henan Provincial Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Czechia (5):
  - RESEARCH SITE s.r.o., Pilsen, Plzeň
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice Olomouc, Pavlov
  - Nemocnice Na Homolce, Prague
  - Krajska zdravotni a.s. - Masarykova nemocnice v Usti nad Labem o.z., Ústí nad Labem
- Poland (6):
  - Beskidzkie Centrum Onkologii im.Jana Pawla II, Bielsko-Biala, Bielsko-Biała
  - LexMedica Osrodek Badan Klinicznych, Wesoła, Weigla
  - KO-MED Centra Kliniczne Biala Podlaska, Biała Podlaska
  - Swietokrzyskie Centrum Onkologii, Kielce
  - Provita Profamilia, Piotrkow Trybunalski
  - Wojewodzki Szpital Specjalistyczny im. J. Korczaka, Słupsk

REFERENCES:
- [Derived] Wang H, Jiang S, Luo H, Zhou F, He D, Ma L, Guo H, Liang C, Chong T, Jiang J, Chen Z, Wang Y, Zou Q, Tian Y, Xiao J, Huang J, Chen J, Dong Q, Zhang X, Li H, Yang X, Lian J, Wang W, Ye D. Patient-reported outcomes of rezvilutamide versus bicalutamide in combination with androgen deprivation therapy in high-volume metastatic hormone-sensitive prostate cancer patients (CHART): a randomized, phase 3 study. Signal Transduct Target Ther. 2024 Dec 18;9(1):351. doi: 10.1038/s41392-024-02064-z. PMID 39690158
- [Derived] Bian X, Gu W, Zhang X, Xie L, Wang S, Shi B, Sun T, Wei S, Weng Z, Xia S, Han B, Xu Z, Xing J, Zhang D, Xu D, Du C, He C, Wang Q, Yang X, Lian J, Wang W, Ye D. Correlation of PSA and survival in metastatic hormone-sensitive prostate cancer treated with rezvilutamide plus ADT in the CHART trial. Med. 2025 Feb 14;6(2):100520. doi: 10.1016/j.medj.2024.09.009. Epub 2024 Oct 16. PMID 39419035
- [Derived] Gu W, Han W, Luo H, Zhou F, He D, Ma L, Guo H, Liang C, Chong T, Jiang J, Chen Z, Wang Y, Zou Q, Tian Y, Xiao J, Huang J, Zhu S, Dong Q, Zhang X, Li H, Yang X, Chen C, Li J, Jin C, Zhang X, Ye D; CHART Investigators. Rezvilutamide versus bicalutamide in combination with androgen-deprivation therapy in patients with high-volume, metastatic, hormone-sensitive prostate cancer (CHART): a randomised, open-label, phase 3 trial. Lancet Oncol. 2022 Oct;23(10):1249-1260. doi: 10.1016/S1470-2045(22)00507-1. Epub 2022 Sep 5. PMID 36075260